CLINICAL TRIAL: NCT06276218
Title: Efficacy of Self - Adjustable Clavicular Brace Versus Standard Clavicular Brace for Treatment of Mid Shaft Clavicle Fracture: A Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Thanachai Klongsangsorn, MD, Prince of Songkla University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PSU
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Clavicle Fracture
Keywords: Clavicle fracture, treatment of clavicle fracture, clavicular brace, figure of eight bandage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-adjustable clavicular brace (Experimental)
  Interventions: Device: Clavicular brace
- standard clavicular brace (Active Comparator)
  Interventions: Device: Clavicular brace

INTERVENTIONS:
Device: Clavicular brace — Clavicular brace for conservative treatment of closed midshaft clavicular fractures

SUMMARY:
A randomized control trial was conducted to compare the outcomes of conservative management for closed midshaft clavicular fractures using self-adjustable clavicular brace and standard clavicular brace.

DETAILED DESCRIPTION:
Ten patients aged 18-75 years with midshaft clavicle fractures were enrolled in the study during February 2022 to February 2023. 6 patients were managed with standard clavicular brace and 4 patients with self-adjustable clavicular brace. All patients were scheduled for follow-up appointments at 1 week, 2 weeks, 4 weeks, 6 weeks and 12 weeks. Results were assessed based on clinical, functional and radiographic outcomes using the DASH questionnaire, pain, measured by VAS, analgesic usage, displacement, shortening, time to union, and patient satisfaction,

ELIGIBILITY:
Inclusion Criteria:

* Patient with aged between 18 - 75 years old
* Closed isolated fracture midshaft of clavicle within 9 days after the injury date

Exclusion Criteria:

* After bracing, fracture displacement and/or shortening > 2 cm or fracture comminution > 3 fragments
* Segmental fracture
* Open fracture
* Impending open fracture (soft tissue compromise/skin lesion)
* Ipsilateral upper extremities fracture which disturbs clavicular bracing
* Floating shoulder which surgical treatment is indicated.
* Patients with other injuries (e.g. head injury, chest and abdomen injury) which interrupted clavicular bracing
* Pathologic fracture
* Patient has limitation for clavicular brace application
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-16 (Estimated)

PRIMARY OUTCOMES:
DASH | 1, 2, 4, 6, 12 week
  DISABILITIES OF THE ARM, SHOULDER AND HAND

SECONDARY OUTCOMES:
Pain, analgesic usage, radiographic outcomes, time to union, and patient satisfaction | 1, 2, 4, 6, 12 week
  Pain, analgesic usage, radiographic outcomes, time to union, and patient satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Songkla University, Songkhla, Hatyai, Thailand

IPD SHARING:
Plan to Share IPD: No